CLINICAL TRIAL: NCT05530408
Title: Quantitative Pulmonary Imaging Registry & Biorepository
Acronym: PIBR
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Peter J. Niedbalski, PhD, Research Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY00148295
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Disease
Keywords: Xenon; Xe-129; CT
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this project is to establish a registry and biorepository of images and biological samples from subjects undergoing novel pulmonary imaging methods to be used for future research aimed toward identifying clinical applications of imaging methods and toward understanding the physiological significance of imaging biomarkers. This registry and biorepository will accelerate the development of these imaging techniques and may lead toward future clinical adoption of quantitative pulmonary imaging.

DETAILED DESCRIPTION:
Imaging is increasingly used for the non-invasive assessment of pulmonary health. Alongside this increased usage, there is enhanced interest in quantitative imaging methods that provide robust, repeatable, and objective measures of lung structure and function. At the forefront of this effort is quantitative computed tomography (qCT). CT imaging is the gold standard for high-resolution imaging of pulmonary structure, and the underlying physics of CT imaging is highly amenable to quantitative analysis.

In addition to qCT, MRI is garnering increased interest as a modality for pulmonary imaging. Like CT, MRI is non-invasive, and it has the additional advantage of being ionizing radiation-free, making it more suitable for repeat imaging and for use in pediatric patients. Traditionally, MRI was not often used for lung imaging due to several difficulties regarding the acquisition of quality images in the lungs. However, recent advances to pulmonary MRI methods have enabled the acquisition of high-quality images of pulmonary structure and function. These advances include the use of ultra-short and zero echo time (UTE and ZTE, respectively) MRI methods, as well as the use of gaseous contrast agents such as hyperpolarized 129Xe.

Despite these advances in qCT and MRI methods, the clinical applications for these imaging techniques are often unclear. Moreover, as new techniques, many of the imaging biomarkers in use have been independently developed by multiple sites and thus require standardization. As such, there is an urgent need both to standardize imaging/analysis techniques and to determine optimal clinical applications for these novel quantitative imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* The participant is enrolling/has enrolled in a research study at the University of Kansas Medical Center that involves Pulmonary MRI and/or Pulmonary CT.

Exclusion Criteria:

* The participant declines to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participating in an Imaging Study at KUMC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Collect Clinical Data | From Enrollment to 3 Months
  Collect relevant medical history (including demographic information, diagnoses, medical tests, smoking history), for patients participating in pulmonary imaging research.
Establish a Biorepository | From Enrollment to 3 Months
  Establish a collection of biospecimens from imaging subjects to foster an improved understanding of the physiological significance of imaging biomarkers.
Biospecimen Collection | From Enrollment to 6 Months
  Correlate imaging biomarkers with biospecimens and physiological/vital signs data.
Collaborate | From Enrollment to 12 Months
  Provide images and biospecimens to researchers working to develop analysis methods for pulmonary CT and MRI. Separate IRB approval, alongside appropriate data and/or materials transfer agreements will be needed for these studies.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Niedbalski, PhD, Principal Investigator — Research Assistant Professor; Luigi R Boccardi, MPH, Study Director — Director of Pulmonary, Critical Care, & Sleep Research
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Collaborators at KUMC that are not on the study team may request access to identified or deidentified data/biospecimens from this project. Collaborators may include parties outside of KUMC, in which case only deidentified data will be shared. When potential collaborators request access to data and/or biospecimens, the following will be considered: research question and study design, timing of request, and amount of specimen needed. Corporate entities will not be allowed access to data or samples from the biobank.
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: Contact Peter J. Niedbalski, PhD to discuss accessing IPD.

REFERENCES:
- See also: KUMC Research - Quantitative Pulmonary Imaging Core — https://www.kumc.edu/school-of-medicine/academics/departments/internal-medicine/divisions/pulmonary-critical-care-and-sleep-medicine/research/quantitative-pulmonary-imaging.html